CLINICAL TRIAL: NCT07332975
Title: A Proportion of ctDNA Positive Patients Diagnosed With cT1bN0 and cT1cN0 TNBC (ARES)
Brief Title: ctDNA Positive Patients Diagnosed With cT1bN0 and cT1cN0 TNBC
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Marija Balic, MD PhD, Professor of Medicine, Hematology Oncology, University of Pittsburgh
Other Study IDs: HCC 25-105
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: ctDNA
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating free DNA (cfDNA); paired tumor and matched WBC whole genome sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This translational biomarker study will collect blood in patients Stage I triple negative breast cancer at diagnosis prior to either neoadjuvant treatment or surgery and then during treatment.

DETAILED DESCRIPTION:
A highly sensitive, tumor-informed method of detecting circulating free DNA (cfDNA) shed by solid tumors has been developed. Plasma will be assayed for ctDNA using the SaferSeqS tumor-informed assay employing DNA sequences derived from breast biopsies and/ or surgery specimens. The abundance and molecular characteristics of ctDNA will be evaluated in 77 patients using optimum Simon Stage II statistical design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 years of age
2. Cytologically or histologically confirmed and previously untreated invasive breast cancer that is:

   * Clinical stage I
   * ≤2 cm on imaging
   * cN0
   * cM0
   * Grade 2 or Grade 3
3. ECOG 0-2
4. Locally assessed ER+ in 0% of cells.
5. Locally assessed HER2-negative (IHC 2+/FISH-negative or IHC 0 or 1+ /either FISH-negative or untested).
6. No prior chemotherapy
7. Fit for chemotherapy and surgery
8. Must have the ability to understand and the willingness to sign a written informed consent document.
9. Must be willing to provide serial blood samples for the study.

Exclusion Criteria:

1. History of other invasive malignancy in the past 2 years
2. Synchronous breast cancers and multifocal/multicentric breast cancers
3. Medical condition or social situation that may preclude adherence to the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage I triple negative breast cancer at diagnosis prior to either neoadjuvant treatment or surgery and then during treatment.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA detection | Up to 2 years
  Detection of ctDNA by assay in blood collected prior to radical prostatectomy using the Vogelstein lab assay. This assay is a highly sensitive, tumor-informed method of detecting circulating free DNA (cfDNA) shed by solid tumors. This assay has shown prognostic value for recurrence and predictive for benefit of adjuvant chemotherapy.

SECONDARY OUTCOMES:
ctDNA clearing | Up to 2 years
  Percentage of patients clearing the ctDNA during neoadjuvant treatment.
pCR rate | Up to 2 years
  pCR rate (ypT0/is) - All mutations per patient tested in one multiplex PCR reaction containing primers for all 96 mutations. This approach allows the detection of as few as one mutant molecule shed from tumor cells into the circulation per hour, and this detection is sufficient to engender high confidence that the patient has residual disease.
ctDNA after surgery treatment | Up to 2 years
  Percentage of patients with ctDNA after surgery and all treatment.
Event free survival (EFS) | Up to 2 years
  Length of time after primary treatment that the patient remains free of related complications or events.
Invasive disease-free survival (IDFS) | Up to 2 years
  Time until the first occurrence of invasive breast cancer recurrence, distant recurrence, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Marija Balic, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No